CLINICAL TRIAL: NCT02100761
Title: Impact of Cytochrome P450 2C19 Genotype Polymorphism on Voriconazole Trough Concentration in Chinese Adult Patients With Invasive Pulmonary Aspergillosis: a Prospective Multicenter Research
Brief Title: CYP 2C19 Polymorphism and Voriconazole Trough Concentration in Chinese Adult Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: dingshifang (Other)
Collaborators: Shandong Provincial Hospital (Other Government); Qianfoshan Hospital (Other); Shandong thorax hospital (Unknown); Jinan Military General Hospital (Other); Jinan Central Hospital (Other)
Responsible Party: Sponsor-Investigator, dingshifang, Professor, Qilu Hospital of Shandong University
Organization: Qilu Hospital of Shandong University (Other)
Other Study IDs: KYLL-2014(KS)-085
Record Dates: First submitted 2014-03-03; First posted 2014-04-01 (Estimated); Last update posted 2014-04-01 (Estimated); Status verified 2014-03

CONDITIONS: Invasive Pulmonary Aspergillosis
Keywords: Voriconazole; Invasive pulmonary aspergillosis; Therapeutic drug monitoring; CYP genetic polymorphism; Efficacy; Safety
MeSH Terms: conditions — Invasive Pulmonary Aspergillosis | interventions — Voriconazole

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — The susceptibility test of aspergillosis strains to voriconazole, serum galactomannan (GM) test, voriconazole trough levels and genotyping of CYP2C19 will be measured.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- invasive pulmonary aspergillosis: Patients with invasive pulmonary aspergillosis and will be treated with voriconazole according to their physician decision in five hospital, Jinan, China
  Interventions: Drug: Voriconazole

INTERVENTIONS:
Drug: Voriconazole — Patients with creatinine clearance at least 50 ml/min will be treated with voriconazole by intravenous drip infusion at the dose of 6 mg/kg twice daily on the first day (Day 1) and 4 mg/kg twice daily from day 2 onward. The IV treatment is at least 7 days. Then switch to 200 mg orally twice daily between meals. The total treatment duration is at least 14 days Patients with creatinine clearance <50 ml/min will be treated with oral voriconazole (loading dose of 400 mg twice daily followed by maintenance dose of 200 mg twice daily between meals for at least 14.0 days).
  Other Names: Voriconazole Intravenous Solution 200 mg; Voriconazole Tablet 50 mg / Voriconazole Tablet 200 mg

SUMMARY:
To investigate the relationship between cytochrome P450 (CYP) 2C19 genetic polymorphism and the steady-state blood concentration of voriconazole in Chinese patients with invasive pulmonary aspergillosis (IPA), and to assess the effects of voriconazole trough concentration on the prognosis of IPA patients.

DETAILED DESCRIPTION:
Each isolate of aspergillosis will be recovered from clinical specimens (sputum, bronchoalveolar lavage fluid, lung biopsy tissue) and the identification of species level will also be performed in Qilu Hospital by using conventional methods (both macroscopic and microscopic characteristics). The aspergillosis strains will be stored in 10 % glycerol broth at -80 °C. The in vitro antifungal susceptibility test of aspergillosis strains to voriconazole will be performed in the Centre for Medical Mycology and Mycoses, First Hospital, Peking University, and the performance will be according to the Clinical and Laboratory Standards Institute (CLSI) standard M38-A2 microdilution methods.

Serum galactomannan (GM) test will be performed twice per week for the first two weeks. A double-sandwich ELISA GM assay was used. A cut-off of optical density index (ODI) >0.5 was taken as positive.

Voriconazole serum levels will be measured on day 4, day 7, day 10, and day 14 (all trough levels). In brief, quantitative analysis of voriconazole was performed using high-performance liquid chromatography coupled with tandem mass spectrometry.

Genotyping of CYP2C19 will be performed using 3 ml of peripheral blood sampled into EDTA (ethylenediaminetetraacetic acid) tubes at day 4. Genomic DNA was extracted from blood leukocytes with the use of a DNA extraction kit. Genotyping was confirmed by polymerase chain reaction (PCR)-restriction fragment length polymorphism (RFLP) analysis. Individuals can be divided into three groups according to the CYP2C19 genotype. Those who inherit two mutant CYP2C19 alleles (*2 and/or *3) have a reduced capacity to metabolize CYP2C19 substrates and are defined as poor metabolizers (PMs). Individuals who are homozygous (*1/*1) for wild-type CYP2C19*1 or 1 wild-type allele and 1 CY¬P2C19*17 have efficient enzymes to metabolize CYP2C19 substrates and are defined as extensive metabolizers (EMs). Subjects who are heterozygous (*1/*2, *1/*3) for wild-type CYP2C19*1 are defined as intermediate metabolizers (IMs)

ELIGIBILITY:
Inclusion Criteria:

* Proven, probable, or possible invasive pulmonary aspergillosis (IPA)
* Acute IPA defined as duration of clinical syndrome of <30 days.
* Treatment with voriconazole
* At least 18 years and older
* Weight >40 kg and ≤120 kg
* Given the informed consent

Exclusion Criteria:

* Patients allergic to azole(s)
* Patients who heve been prescribed voriconazole before
* Positive urine pregnancy test (if female)
* Patients with aspergilloma or chronic aspergillosis ( >1 month duration )
* Anticipated survival of less than 5 days or Karnofsky score <=20

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with invasive pulmonary aspergillosis and will be treated with voriconazole according to their physician decision
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2014-06; Primary Completion 2015-06 (Estimated); Study Completion 2015-06 (Estimated)

PRIMARY OUTCOMES:
voriconazole trough level | one year

SECONDARY OUTCOMES:
Overall mortality | one year

CONTACTS AND LOCATIONS:
Overall Officials: Shifang Ding, Ph.D., Study Chair — Qilu Hospital of Shandong University
Locations (1):
- Qilu Hospital, Jinan, Shandong, China